CLINICAL TRIAL: NCT00631969
Title: Pivotal Phase III Trial to Investigate the Efficacy and Safety of an Orodispersible Tablet Vardenafil Versus Placebo in the Treatment of Men With Erectile Dysfunction (ED) - a Fixed-dose, Double-blind, Randomized Multi-center Trial - POTENT I
Brief Title: Vardenafil ODT Versus Placebo in Males With Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12093; 2008-000536-40 (EudraCT Number)
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vardenafil ODT (STAXYN, BAY38-9456) (Experimental): Vardenafil 10 mg orodispersible tablet (ODT) taken on demand (PRN), approximately one hour before start of sexual activity, no more than one dose per day.
  Interventions: Drug: Vardenafil ODT (STAXYN, BAY38-9456)
- Placebo (Placebo Comparator): Matching placebo tablet taken on demand (PRN), approximately one hour before start of sexual activity, no more than one dose per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vardenafil ODT (STAXYN, BAY38-9456) — Subjects will receive 12 weeks of PRN (on demand) treatment with Vardenafil 10mg orodispersible tablet (ODT)
  Arms: Vardenafil ODT (STAXYN, BAY38-9456)
Drug: Placebo — Subjects will receive 12 weeks of PRN (on demand) treatment with matching placebo tablet
  Arms: Placebo

SUMMARY:
This study investigates the safety and efficacy of a new dosage form of Vardenafil, an orodispersible tablet (ODT), and compares it to the safety and efficacy of a placebo (inactive) tablet in the treatment of erectile dysfunction. After a 4-week unmedicated phase, patients will receive Vardenafil ODT or matching placebo for 12 weeks. Safety will be determined by laboratory and other evaluations. Efficacy will be determined by the results of different questionnaires and the patient diary that will be used.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 years-of-age or older
* Stable, heterosexual relationship for at least 6 months
* A history of erectile dysfunction (ED) for at least 6 months

Exclusion Criteria:

* Any underlying cardiovascular condition, including unstable angina pectoris
* History of myocardial infarction, stroke or life-threatening arrhythmia within 6 months prior to visit 1
* Uncontrolled atrial fibrillation / flutter at screening
* History of surgical prostatectomy for prostate cancer
* Hereditary degenerative retinal disorders
* History of loss of vision because of Non-arteritic anterior ischemic optic neuropathy (NAION), temporary or permanent loss of vision
* Presence of penile anatomical abnormalities
* Subjects who have been confirmed with phenylketonuria (PKU)
* Spinal cord injury
* Resting or postural hypotension or hypertension
* Subjects who are taking nitrates or nitric oxide donors, androgens, anti-androgens, alpha- blockers, medication known to prolong QT interval, Human immunodeficiency virus (HIV) protease inhibitors, itraconazole or ketoconazole, an clarithromycin and erythromycin
* Use of any treatment for ED within 7 days of Visit 1
* History of congenital QT prolongation
* History of syncope within the last 6 months prior to entry into the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (36):
- Belgium (5):
  - Antwerp
  - Bruxelles - Brussel
  - Genk
  - Ghent
  - Liège
- France (5):
  - Lille
  - Lyon
  - Marseille
  - Mont-de-Marsan
  - Paris
- Germany (9):
  - München, Bavaria
  - Weiden, Bavaria
  - Hamburg, Hamburg
  - Osnabrück, Lower Saxony
  - Mönchengladbach, North Rhine-Westphalia
  - Mülheim, North Rhine-Westphalia
  - Bautzen, Saxony
  - Leipzig, Saxony
  - Meissen, Saxony
- Netherlands (6):
  - Arnhem
  - Deurne
  - Leiden
  - Losser
  - Maastricht
  - Nijverdal
- South Africa (6):
  - Centurion, Gauteng
  - Johannesburg, Gauteng
  - Krugersdorp, Gauteng
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
- Spain (5):
  - Alicante, Alicante
  - Barcelona, Barcelona
  - San Cristóbal de La Laguna, La Laguna
  - Valencia, Valencia
  - Vigo, Vigo

REFERENCES:
- [Result] Debruyne FM, Gittelman M, Sperling H, Borner M, Beneke M. Time to onset of action of vardenafil: a retrospective analysis of the pivotal trials for the orodispersible and film-coated tablet formulations. J Sex Med. 2011 Oct;8(10):2912-23. doi: 10.1111/j.1743-6109.2011.02462.x. Epub 2011 Aug 30. PMID 21883954
- [Result] Sperling H, Debruyne F, Boermans A, Beneke M, Ulbrich E, Ewald S. The POTENT I randomized trial: efficacy and safety of an orodispersible vardenafil formulation for the treatment of erectile dysfunction. J Sex Med. 2010 Apr;7(4 Pt 1):1497-507. doi: 10.1111/j.1743-6109.2010.01806.x. Epub 2010 Mar 3. PMID 20233275
- [Result] Heinig R, Weimann B, Dietrich H, Bottcher MF. Pharmacokinetics of a new orodispersible tablet formulation of vardenafil: results of three clinical trials. Clin Drug Investig. 2011;31(1):27-41. doi: 10.2165/11584950-000000000-00000. PMID 20925442
- [Result] Sperling H, Gittelman M, Norenberg C, Ulbrich E, Ewald S. Efficacy and safety of an orodispersible vardenafil formulation for the treatment of erectile dysfunction in elderly men and those with underlying conditions: an integrated analysis of two pivotal trials. J Sex Med. 2011 Jan;8(1):261-71. doi: 10.1111/j.1743-6109.2010.02005.x. Epub 2010 Aug 30. PMID 20807322
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited to 40 investigational centers in Belgium (4), France (8), Germany (9), Spain (3), Netherlands (5), and South Africa (11). First patient first visit on 25 April 2008, last patient last visit on 19 January 2009.
Pre-assignment Details: 409 male subjects screened (<65 years: n=185; >=65 years: n=224), 362 randomized to treatment (186 to Vardenafil ODT, and 176 to placebo). The main efficacy analysis set was the Intent-to-treat (ITT) population (randomized treated subjects with baseline and post-baseline efficacy and safety assessments); 183 on Vardenafil ODT and 172 on placebo.
Period: Overall Study
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Started | 186 | 176
Received Treatment | 184 (safety population) | 174 (safety population)
Completed | 171 | 155
Not Completed | 15 | 21
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 2 | 8
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Consent Withdrawn | 5 | 7
Not completed — Noncompliant With Study Medication | 0 | 1
Not completed — No Drug Exposure | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo | Total
Number analyzed (Participants) | 184 | 174 | 358
Age, Customized [Number; unit: Participants]
  <65 years | 87 | 81 | 168
  >=65 years | 97 | 93 | 190
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 184 | 174 | 358
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms per square meter (kg/m^2)]
  All age groups | 27.2 (3.4) | 27.5 (4.0) | 27.3 (3.7)
  < 65 years | 27.5 (3.5) | 27.9 (4.3) | 27.7 (3.9)
  >= 65 years | 26.9 (3.2) | 27.1 (3.6) | 27.0 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Index of Erectile Function (IIEF-EF Sub-Score) at 12 Weeks or LOCF
Description: The primary variable was the treatment group difference from baseline to Week 12 or Last observation carried forward (LOCF) of the least square mean difference in the IIEF-EF domain score (1-30 ordinal points, specifying the severity of erectile dysfunction: <=10 'severe'; 11-16 'moderate'; 17-21 'mild to moderate'; 22-25 'mild'; >25 'no ED').
Time Frame: from baseline up to 12 weeks
Population: The primary data set was the ITT (Intent-to treat) population defined as all randomized treated subjects with baseline and post-baseline efficacy data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 183 | 172
scores on a scale
  <65 years | 9.6 (6.28) | 2.1 (7.33)
  ≥65 years | 7.7 (8.19) | 0.9 (6.42)
  Total | 8.6 (7.40) | 1.4 (6.86)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Power adjustment for 3 primary efficacy variables (3 variables have to be significant in favor of Vardenafil to conclude efficacy). Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -7.109, 95% CI [-8.562 to -5.6561]

2. Primary Outcome: Change in Percentage From Baseline in Success of Penetration at 12 Weeks
Description: Sexual encounter profile (SEP) items success rates are the percentage of all valid and successful intercourse attempts (items answered 'yes') in relation to all valid attempts. Here the SEP item refers to the ability to penetrate the partner.
Time Frame: from baseline up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of successful penetrations
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 179 | 169
percentage of successful penetrations
  <65 years | 35.8 (33.63) | 5.5 (42.82)
  ≥65 years | 35.2 (38.06) | 8.7 (28.41)
  Total | 35.5 (35.93) | 7.2 (35.79)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -29.027, 95% CI [-35.519 to -22.534]

3. Primary Outcome: Change From Baseline in Success of Erection Maintenance at 12 Weeks
Description: SEP items success rates are the percentage of all valid and successful intercourse attempts (items answered 'yes') in relation to all valid attempts. Here the SEP item refers to the ability to maintain an erection after penetration.
Time Frame: from baseline up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of success in maintenance
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 178 | 164
percentage of success in maintenance
  <65 years | 54.5 (32.72) | 15.2 (31.30)
  ≥65 years | 49.2 (37.28) | 7.7 (25.72)
  Total | 51.7 (35.18) | 11.3 (28.67)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -38.193, 95% CI [-45.021 to -31.366]

4. Secondary Outcome: Percentage of Subjects Achieving "Back to Normal" Erectile Function
Description: Responders: percentage of subjects achieving an IIEF-EF score > 25. The primary variable was the treatment group difference from baseline to Week 12 or Last observation carried forward (LOCF) of the least square mean difference in the IIEF-EF domain score (1-30 ordinal points, specifying the severity of erectile dysfunction: <=10 'severe'; 11-16 'moderate'; 17-21 'mild to moderate'; 22-25 'mild'; >25 'no ED').
Time Frame: up to 12 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 181 | 172
percentage of participants
  <65 years | 46 | 13
  ≥65 years | 34 | 11
  Total | 40 | 12
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) adjusted for age group and pooled center; Cochran-Mantel-Haenszel = 34.778

5. Secondary Outcome: Change in Percentage From Baseline in Ability to Obtain an Erection at 12 Weeks
Description: SEP items success rates are the percentage of all valid and successful intercourse attempts (items answered 'yes') in relation to all valid attempts. Here the SEP item refers to the ability to obtain successful erections.
Time Frame: from baseline up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of successful erections
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 180 | 169
percentage of successful erections
  <65 years | 18.8 (29.6) | -1.8 (37.86)
  ≥65 years | 14.6 (33.21) | 1.2 (37.43)
  Total | 16.6 (31.54) | -0.2 (37.55)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -16.503, 95% CI [-22.424 to -10.764]

6. Secondary Outcome: Change in Percentage From Baseline in Satisfaction With the Hardness of Erection at 12 Weeks
Description: SEP items success rates are the percentage of all valid and successful intercourse attempts (items answered 'yes') in relation to all valid attempts. Here the SEP item refers to the ability to get satisfactory hardness of erections.
Time Frame: from baseline up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of satisfactory erections
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 179 | 164
percentage of satisfactory erections
  <65 years | 51.7 (36.10) | 11.2 (27.69)
  ≥65 years | 45.3 (43.09) | 7.5 (27.70)
  Total | 48.4 (39.95) | 9.2 (27.67)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -38.167, 95% CI [-45.261 to -31.073]

7. Secondary Outcome: Change in Percentage From Baseline in Overall Satisfaction at 12 Weeks
Description: SEP items success rates are the percentage of all valid and successful intercourse attempts (items answered 'yes') in relation to all valid attempts. Here the SEP item refers to overall satisfactory attempts.
Time Frame: from baseline up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of satisfactory attempts
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 178 | 164
percentage of satisfactory attempts
  <65 years | 55.7 (36.83) | 14.4 (30.26)
  ≥65 years | 45.8 (38.43) | 5.6 (25.74)
  Total | 50.5 (37.90) | 9.8 (28.24)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -36.555, 95% CI [-43.645 to -29.465]

8. Secondary Outcome: Change in Percentage From Baseline in Ability to Ejaculate at 12 Weeks
Description: SEP items success rates are the percentage of all valid and successful intercourse attempts (items answered 'yes') in relation to all valid attempts. Here the SEP item refers to the ability to have successful ejaculations.
Time Frame: from baseline up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of ejaculation successes
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 179 | 163
percentage of ejaculation successes
  <65 years | 34.5 (36.19) | 5.4 (36.86)
  ≥65 years | 32.7 (35.23) | 10.1 (29.96)
  Total | 33.5 (35.60) | 7.9 (33.38)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -25.193, 95% CI [-31.562 to -18.824]

9. Secondary Outcome: Number of Sexual Attempts Till First Successful Attempt
Time Frame: up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Sexual Attempts
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 180 | 169
Sexual Attempts
  <65 years | 1.0 (2.6) | 2.7 (4.4)
  ≥65 years | 1.4 (3.1) | 4.4 (7.4)
  Total | 1.2 (2.9) | 3.6 (6.2)

10. Secondary Outcome: Change From Baseline in Ease With Erection at 12 Weeks or LOCF
Description: Treatment group difference in points on the Treatment Satisfaction Scale (TSS, 0-100 normalized ordinal scores, higher scores indicate greater levels of 'ease with erection', 'erectile functioning satisfaction', 'pleasure of sexual activity', 'satisfaction with orgasm', 'confidence for completion', and 'satisfaction with medication') domain "Ease with Erection" from baseline to Week 12 or LOCF expressed as the least square mean difference.
Time Frame: from baseline up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 180 | 168
scores on a scale
  <65 years | 28.6 (28.02) | 4.2 (27.92)
  ≥65 years | 25.0 (31.20) | 0.8 (28.98)
  Total | 26.7 (29.73) | 2.4 (28.46)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -24.703, 95% CI [-30.067 to -19.340]

11. Secondary Outcome: Change From Baseline in Erectile Function Satisfaction at 12 Weeks or LOCF
Description: Treatment group difference in points on the Treatment Satisfaction Scale (TSS, 0-100 normalized ordinal scores, higher scores indicate greater levels of 'ease with erection', 'erectile functioning satisfaction', 'pleasure of sexual activity', 'satisfaction with orgasm', 'confidence for completion', and 'satisfaction with medication') domain " Erectile function satisfaction" from baseline to Week 12 or LOCF expressed as the least square mean difference.
Time Frame: from baseline up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 180 | 168
scores on a scale
  <65 years | 1.3 (1.28) | 0.1 (1.35)
  ≥65 years | 1.2 (1.18) | -0.1 (1.28)
  Total | 1.3 (1.23) | 0.0 (1.31)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -24.496, 95% CI [-34.865 to -24.128]

12. Secondary Outcome: Change From Baseline in Pleasure of Sexual Activity at 12 Weeks or LOCF
Description: Treatment group difference in points on the Treatment Satisfaction Scale (TSS, 0-100 normalized ordinal scores, higher scores indicate greater levels of 'ease with erection', 'erectile functioning satisfaction', 'pleasure of sexual activity', 'satisfaction with orgasm', 'confidence for completion', and 'satisfaction with medication') domain " Pleasure of sexual activity" from baseline to Week 12 or LOCF expressed as the least square mean difference.
Time Frame: from baseline up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 180 | 168
scores on a scale
  <65 years | 28.6 (29.34) | 3.2 (29.06)
  ≥65 years | 25.3 (30.24) | -3.6 (29.48)
  Total | 26.8 (29.78) | -0.4 (29.40)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -27.775, 95% CI [-33.155 to -22.394]

13. Secondary Outcome: Change From Baseline in Satisfaction With Orgasm at 12 Weeks or LOCF
Description: Treatment group difference in points on the Treatment Satisfaction Scale (TSS, 0-100 normalized ordinal scores, higher scores indicate greater levels of 'ease with erection', 'erectile functioning satisfaction', 'pleasure of sexual activity', 'satisfaction with orgasm', 'confidence for completion', and 'satisfaction with medication') domain "Satisfaction with orgasm" from baseline to Week 12 or LOCF expressed as the least square mean difference.
Time Frame: from baseline up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 180 | 168
scores on a scale
  <65 years | 31.0 (29.46) | 7.1 (32.66)
  ≥65 years | 26.8 (32.29) | 5.5 (31.80)
  Total | 28.8 (30.98) | 6.3 (32.11)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -23.326, 95% CI [-29.062 to -17.598]

14. Secondary Outcome: Change From Baseline in Confidence for Completion at 12 Weeks or LOCF
Description: Treatment group difference in points on the Treatment Satisfaction Scale (TSS, 0-100 normalized ordinal scores, higher scores indicate greater levels of 'ease with erection', 'erectile functioning satisfaction', 'pleasure of sexual activity', 'satisfaction with orgasm', 'confidence for completion', and 'satisfaction with medication') domain "Confidence for completion" from baseline to Week 12 or LOCF expressed as the least square mean difference.
Time Frame: from baseline up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 180 | 168
scores on a scale
  <65 years | 28.7 (27.56) | 5.0 (27.53)
  ≥65 years | 25.8 (30.18) | 3.6 (26.57)
  Total | 27.7 (28.94) | 4.2 (26.94)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -23.384, 95% CI [-28.594 to -18.175]

15. Secondary Outcome: Satisfaction With Medication at Week 12 or LOCF
Description: Treatment group difference in points on the Treatment Satisfaction Scale (TSS, 0-100 normalized ordinal scores, higher scores indicate greater levels of 'ease with erection', 'erectile functioning satisfaction', 'pleasure of sexual activity', 'satisfaction with orgasm', 'confidence for completion', and 'satisfaction with medication') domain "Satisfaction with medication" at LOCF expressed as the least square mean difference.
Time Frame: up to 12 weeks
Population: The primary data set was the ITT (Intent-to treat) population defined as all randomized treated subjects with LOCF values.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 180 | 167
scores on a scale
  <65 years | 57.2 (28.09) | 22.1 (25.58)
  ≥65 years | 52.3 (29.54) | 20.4 (24.55)
  Total | 54.6 (28.90) | 21.2 (24.96)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -33.076, 95% CI [-38.745 to -27.407]

16. Secondary Outcome: Patient Self Reported Improvement of Erectile Function Under Treatment Using a Categorical Rating Scale
Description: Categorical Rating Scale is a binary rating scale with 2 response options which is 'yes/no'; percentage of participants with positive answers to the Global Assessment Question. Global Assessment Question (GAQ): 'Has the treatment you have been taking over the past for weeks improved your erection?' (yes/no)
Time Frame: up to 12 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 180 | 168
percentage of participants
  <65 years | 76 | 30
  ≥65 years | 69 | 22
  Total | 72 | 26
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) adjusted for pooled centers and age group; Cochran-Mantel-Haenszel = 74.449

17. Secondary Outcome: Pharmacokinetics Measured as Area Under Curve (AUC) of Vardenafil in Plasma
Description: Plasma concentrations after single dose administration of 10 mg Vardenafil ODT followed for up to 24 hours post-dose.
Time Frame: Visit 5 after 12 weeks of treatment
Population: Pharmacokinetics (PK) were studied in a sub-group of 25 ED patients receiving a single dose of 10 mg Vardenafil ODT on a separate visit. This sub-population comprised 12 patients aged 18-64 years and 13 patients aged 65 years and above. The PK data of one elderly patient were only evaluable for Cmax but not for AUC.
Measure: Geometric Mean (Full Range); unit: μg*h/L
Groups:
- ED Patients Aged < 65 Years: Vardenafil 10 mg orodispersible tablets (ODT) taken on demand (PRN) 1 hour before sexual activity for ED patients aged < 65 years.
- ED Patients Aged ≥ 65 Years: Vardenafil 10 mg orodispersible tablets (ODT) taken on demand (PRN) 1 hour before sexual activity for ED patients aged ≥ 65 years.
Arm/Group | ED Patients Aged < 65 Years | ED Patients Aged ≥ 65 Years
Number analyzed (Participants) | 12 | 12
μg*h/L | 47.16 [18.97 to 112.8] | 55.37 [21.23 to 104.4]
Statistical Analysis 1: Comparison: ED Patients Aged < 65 Years vs ED Patients Aged ≥ 65 Years; Point estimate and 90% confidence interval of ratio (patients aged ≥ 65 years / patients aged < 65 years) were calculated; Test type: Non-Inferiority or Equivalence — This is an exploratory analysis of Vardenafil exposure in ED patients of different age categories to assess the effect of age on the drug's pharmacokinetics; Point estimate of ratio = 117.42, 90% CI [79.59 to 173.23]
Statistical Analysis 2: Comparison: ED Patients Aged < 65 Years vs ED Patients Aged ≥ 65 Years; A linear regression line is fitted to the logarithm of AUC. Test of the hypothesis of a zero slope using the two-sided t-test at α = 0.05; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 17, analysis 1]; p = 0.7064, Regression, Linear

18. Secondary Outcome: Pharmacokinetics Measured as Maximum Concentration (Cmax) of Vardenafil in Plasma
Description: Plasma concentrations after single dose administration of 10 mg Vardenafil ODT followed for up to 24 hours post-dose.
Time Frame: Visit 5 after 12 weeks of treatment
Population: Pharmacokinetics were studied in a sub-group of 25 ED patients receiving a single dose of 10 mg Vardenafil ODT on a separate visit. This sub-population comprised 12 patients aged 18-64 years and 13 patients aged 65 years and above.
Measure: Geometric Mean (Full Range); unit: μg/L
Arm/Group | ED Patients Aged < 65 Years | ED Patients Aged ≥ 65 Years
Number analyzed (Participants) | 12 | 13
μg/L | 10.09 [3.134 to 19.04] | 13.43 [2.913 to 27.91]
Statistical Analysis 1: Comparison: ED Patients Aged < 65 Years vs ED Patients Aged ≥ 65 Years; [analysis description as in outcome 17, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 17, analysis 1]; Point estimate of ratio = 133.07, 90% CI [87.46 to 202.46]
Statistical Analysis 2: Comparison: ED Patients Aged < 65 Years vs ED Patients Aged ≥ 65 Years; A linear regression line is fitted to the logarithm of Cmax. Test of the hypothesis of a zero slope using the two-sided t-test at α=0.05; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 17, analysis 1]; p = 0.8749, Regression, Linear

19. Secondary Outcome: Pharmacokinetics Measured as Area Under Curve (AUC) of Metabolite M-1 (BAY44-5576) in Plasma
Description: Plasma concentrations after single dose administration of 10 mg Vardenafil ODT followed for up to 24 hours post-dose.
Time Frame: Visit 5 after 12 weeks of treatment
Population: Pharmacokinetics were studied in a sub-group of 25 ED patients receiving a single dose of 10 mg Vardenafil ODT on a separate visit. This sub-population comprised 12 patients aged 18-64 years and 13 patients aged 65 years and above. AUC data were not available in 3 elderly patients.
Measure: Geometric Mean (Full Range); unit: µg*h/L
Arm/Group | ED Patients Aged < 65 Years | ED Patients Aged ≥ 65 Years
Number analyzed (Participants) | 12 | 10
µg*h/L | 33.36 [10.94 to 68.46] | 41.80 [16.56 to 148.5]
Statistical Analysis 1: Comparison: ED Patients Aged < 65 Years vs ED Patients Aged ≥ 65 Years; Point estimate and 90% confidence interval of ratio (patients aged ≥ 65 years/ patients aged < 65 years) were calculated; Test type: Non-Inferiority or Equivalence — This is an exploratory analysis of metabolite M-1 exposure in ED patients of different age categories to assess the effect of age on the drug's pharmacokinetics; Point estimate of ratio = 125.28, 90% CI [73.65 to 213.11]
Statistical Analysis 2: Comparison: ED Patients Aged < 65 Years vs ED Patients Aged ≥ 65 Years; A linear regression line is fitted to the logarithm of AUC. Test of the hypothesis of a zero slope using the two-sided t-test at α=0.05; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; p = 0.7375, Regression, Linear

20. Secondary Outcome: Pharmacokinetics Measured as Maximum Concentration (Cmax) of Metabolite M-1 (BAY44-5576) in Plasma
Description: Plasma concentrations after single dose administration of 10 mg Vardenafil ODT followed for up to 24 hours post-dose.
Time Frame: Visit 5 after 12 weeks of treatment
Population: as for outcome 18
Measure: Geometric Mean (Full Range); unit: µg/L
Arm/Group | ED Patients Aged < 65 Years | ED Patients Aged ≥ 65 Years
Number analyzed (Participants) | 12 | 13
µg/L | 9.260 [3.756 to 23.32] | 11.47 [5.563 to 41.17]
Statistical Analysis 1: Comparison: ED Patients Aged < 65 Years vs ED Patients Aged ≥ 65 Years; [analysis description as in outcome 17, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; Point estimate of ratio = 123.84, 90% CI [80.12 to 191.42]
Statistical Analysis 2: Comparison: ED Patients Aged < 65 Years vs ED Patients Aged ≥ 65 Years; A linear regression line is fitted to the logarithm of Cmax. Test of the hypothesis of a zero slope using the two-sided t-test at α = 0.05; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; p = 0.3940, Regression, Linear

ADVERSE EVENTS:
Groups:
- Vardenafil ODT (STAXYN, BAY 38-9456): Vardenafil 10 mg orodispersible tablet (ODT) taken on demand (PRN), approximately one hour before start of sexual activity, no more than one dose per day.
Arm/Group | Vardenafil ODT (STAXYN, BAY 38-9456) | Placebo
Serious Adverse Events (participants affected / at risk) | 4/184 | 1/174
Other Adverse Events (participants affected / at risk) | 70/184 | 36/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vardenafil ODT (STAXYN, BAY 38-9456) (N=184) | Placebo (N=174)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vardenafil ODT (STAXYN, BAY 38-9456) (N=184) | Placebo (N=174)
Angina pectoris (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 1
Bundle branch block right (Cardiac disorders) | 0 | 3
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Supraventricular extrasystoles (Cardiac disorders) | 3 | 2
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Eye disorder (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 7 | 0
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Feeling hot (General disorders) | 2 | 0
Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Sluggishness (General disorders) | 0 | 1
Induration (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 30 | 2
Memory impairment (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Pharmaceutical product complaint (Social circumstances) | 0 | 3
Meniscus removal (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1
Flushing (Vascular disorders) | 14 | 0
Hypertension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the protocol it is specified that all results are the property of the sponsor. The investigator must discuss any publication with the sponsor prior to release and obtain written consent of the sponsor. The investigator must send a draft publication to the sponsor thirty days in advance of submission in order to obtain approval prior to submission of the final version for publication.